CLINICAL TRIAL: NCT01012778
Title: Implementation of a Multimodal Program Including Yoga and Meditation as Well as Play Therapy for ADHD and Dyslexia in a Public School in Najibabad, India
Brief Title: Implementation of Climb Up Program for Children With Attention Deficit Hyperactivity Disorder (ADHD) and Dyslexia in a School in India
Acronym: ClimbUp
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Climb Up Kids (Other)
Responsible Party: Principal Investigator, Devendra I Mehta, PI, Climb Up Kids
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAJMDKV2007
Record Dates: First submitted 2009-11-05; First posted 2009-11-13 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Attention Deficit Hyperactivity Disorder; Dyslexia
Keywords: Performance impairment; Yoga; Meditation; Peer mediated
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Dyslexia

ARMS (1):
- Climbup ADHD and Dyslexia Program (Experimental): Open label - intervention with pre and post parameters collected
  Intervention: Yoga, Meditation, Play therapy for children with ADHD and Dyslexia twice a week in classroom with 6 week and 12 month, primary outcomes in terms of Vanderbilt ADHD scores
  Interventions: Behavioral: Climb Up ADHD and Dyslexia Program

INTERVENTIONS:
Behavioral: Climb Up ADHD and Dyslexia Program — Using a peer mediated multimodal intervention program for ADHD and Dyslexia use Yoga, Meditation, Play therapy administered by (trained) high school volunteers

SUMMARY:
A multimodal intervention was rolled out at a large public school in Najibabad, Uttar Pradesh (UP). The program identified elementary school children with ADHD and Dyslexia using standard screening of all children who had performance impairment in at least one domain of the Vanderbilt questionnaire. The program consisted of play therapy, physical exercise, yoga and meditation. The program was established by High school volunteers from The US and UK over 6 weeks. Once implemented during the morning of school, high school volunteers from the school were trained to continue the program. Vanderbilt questionnaires were completed at intervals to allow follow up.

ELIGIBILITY:
Inclusion Criteria:

* All children between 6 and 11 years attending MDKV public school in Najibabad, UP who had assessment performed for ADHD or Dyslexia

Exclusion Criteria:

* Children who were not enrolled by the parents

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2007-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Changes in ADHD scores using Vanderbilt | Intervals of 6 months

SECONDARY OUTCOMES:
Improvement in self-care as assessed by improvement in dental Decayed, Missing and Filled Teeth (DMFT) scores | 6 to 12 month interval changes
Improvement in speed and accuracy of reading samples for children with Dyslexia | 6 to 12 monthly

CONTACTS AND LOCATIONS:
Overall Officials: Devendra Mehta, MBBS MSC MRCP, Principal Investigator — Arnold Palmer Hospital for Children
Locations (1):
- MDKV Schools, Najībābād, Uttar Pradesh, India